CLINICAL TRIAL: NCT01753154
Title: The Effect of Balance PD Solution on the Peritoneal Membrane in Patients on Automated Peritoneal Dialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PD-NL-04-EU
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Renal Failure
Keywords: Peritoneal Dialysis; Biocompatible dialysis solution; Hydration status; Residual renal function; Body composition monitor; Bioimpedance spectroscopy; Cancer antigen 125
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Solution B (balance PD solution) (Experimental): Treatment 8 weeks with solution B (balance PD solution), next 8 weeks with solution A (conventional PD solution)
  Interventions: Drug: Solution B (balance PD solution)
- Solution A (conventional PD solution) (Active Comparator): Treatment 8 weeks with solution A (conventional PD solution), next 8 weeks with solution B (balance PD solution)
  Interventions: Drug: Solution A (conventional PD solution)

INTERVENTIONS:
Drug: Solution B (balance PD solution) — balance 1.5% glucose, solution for peritoneal dialysis; balance 2.3% glucose, solution for peritoneal dialysis; balance 4.25% glucose, solution for peritoneal dialysis, each with 1.25 mmol/l or 1.75 mmol/l calcium
  Other Names: Balance
  Arms: Solution B (balance PD solution)
Drug: Solution A (conventional PD solution) — Solutions for peritoneal dialysis: CAPD 2 (1.5% glucose, 1.75mmmol/l calcium), CAPD 3 (4.25 % glucose, 1.75mmmol/l calcium), CAPD 4 (2.3% glucose, 1.75mmmol/l calcium), CAPD 17 (1.5% glucose, 1.25mmmol/l calcium), CAPD 18 (4.25% glucose, 1.25mmmol/l calcium) and CAPD 19 (2.3% glucose, 1.25mmmol/l calcium)
  Other Names: CAPD 2, CAPD 3, CAPD 4, CAPD 17, CAPD 18 and CAPD 19
  Arms: Solution A (conventional PD solution)

SUMMARY:
To investigate the biocompatibility of the peritoneal dialysis (PD) solution balance in comparison to the conventional PD solution in APD(automated peritoneal dialysis) patients using the APD cycler sleep•safe.

DETAILED DESCRIPTION:
Equivalence of the investigational PD solution balance regarding fluid status compared to the conventional PD solution.

Effects of balance on inflammation and systemic advanced glycation end products formation.

Effects of balance on peritoneal and total urea clearance, on peritoneal and total creatinine clearance and on ultrafiltration, on residual diuresis and on cholesterol levels.

Safety of the investigational PD solution balance and the conventional PD solution as a control drug.

The mesothelial cell mass assessed by Cancer Antigen 125 is affected by the use of the type of PD solution in APD patients using sleep•safe. Treating patients with the PD solution balance leads to not more than 1 litre difference in hydration in comparison to the conventional PD solution which is considered as clinically not relevant regarding blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* APD patient ≥ 18 years
* Prevalent patient with at least 3 months experience on APD prior to inclusion
* Patient is trained on and being treated with the sleep•safe APD cycler
* Patient treated on APD exclusively with registered conventional PD solutions CAPD 2, CAPD 3, CAPD 4, CAPD 17, CAPD 18 or CAPD 19 for at least 8 weeks prior to inclusion
* Patient is on stable diuretic treatment e.g no change in diuretic treatment within the last 30 days prior to inclusion
* Informed consent signed and dated by study patient and investigator/authorised physician
* Ability to understand the nature and requirements of the study

Exclusion Criteria:

* Peritonitis treatment £ 4 weeks preceding inclusion
* APD patients treated with IPD modality (intermittent peritoneal dialysis)
* Malignant disease without remission
* Patients with artificial joints, amputations, stents, or pacemaker
* Patients with congestive heart failure or coronary artery disease NYHA (New York Heart Association) III and higher
* Active HBV (hepatitis B virus)or HCV(hepatitis C virus)infection- HIV positive
* Participation in an interventional clinical study during the preceding 30 days
* Any condition which could interfere with the patient's ability to comply with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
CA 125 (cancer antigen 125) appearance rate in the 24 hours effluent and estimated hydration | 16 weeks
  The appearance rate is defined as the sum of the amount of CA125 determined in each outflow bag (concentration of CA125 in outflow multiplied with outflow volume) divided by the real cumulative dwell time of all dwells performed on the day of the 24-hour dialysate collection.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Feriani, MD, Principal Investigator — Ospedale Umberto Oo, 30174 Mestre, Italy
Locations (7):
- Poland (3):
  - Centrum Dializ Fresenius Nephrocare, Gdansk
  - Uniwersytecki Szpital Kliniczny nr 1, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin
- Spain (4):
  - Complejo hospitalario universitario de Albacete, Albacete
  - Fundación Hospital Alcorcón, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid